CLINICAL TRIAL: NCT00047281
Title: Trial Of Oral Thalidomide, Celecoxib, Etoposide And Cyclophosphamide In Adult Patients With Relapsed Or Progressive Malignant Gliomas
Brief Title: Thalidomide, Celecoxib, and Combination Chemotherapy in Treating Patients With Relapsed or Refractory Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Schering-Plough (Industry); Celgene (Industry)
Responsible Party: Principal Investigator, Patrick Y. Wen, MD, Director, Center for Neuro-Oncology, Dana-Farber Cancer Institute
Masking: None | Purpose: Treatment
Other Study IDs: 01-278; P30CA006516 (NIH); CDR0000257584; NCI-G02-2117; CELGENE-2001-P-001757/3
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult glioblastoma; adult mixed glioma; recurrent adult brain tumor; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Glioblastoma; Glioma; Brain Neoplasms; Gliosarcoma | interventions — Celecoxib; Cyclophosphamide; Etoposide; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: celecoxib
Drug: cyclophosphamide
Drug: etoposide
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide and celecoxib may stop the growth of tumor cells by stopping blood flow to the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining thalidomide and celecoxib with etoposide and cyclophosphamide may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining thalidomide and celecoxib with etoposide and cyclophosphamide in treating patients who have relapsed or refractory malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of thalidomide, celecoxib, etoposide, and cyclophosphamide, in terms of 6-month progression-free survival, in patients with relapsed or refractory malignant glioma.
* Determine the overall survival of patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine the radiographic response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral thalidomide once daily and oral celecoxib twice daily on days 1-42, oral etoposide once daily on days 1-21, and oral cyclophosphamide once daily on days 22-42. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 48 patients (32 with glioblastoma multiforme and 16 with anaplastic glioma) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed intracranial malignant glioma, including glioblastoma multiforme, gliosarcoma, anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic mixed oligoastrocytoma, or malignant astrocytoma not otherwise specified
* Unequivocal evidence of relapsed or refractory disease by MRI or CT scan and/or tumor resection

  * Steroid therapy prior to MRI or CT scan must have been at a stable dose for at least 5 days
  * Failed prior radiotherapy

    * Must have confirmation of true progression rather than radiation necrosis if previously treated with interstitial brachytherapy or stereotactic radiosurgery

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* More than 2 months

Hematopoietic

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin greater than 9 g/dL
* No history of bleeding disorder

Hepatic

* Bilirubin less than 1.5 mg/dL
* SGPT less than 2.5 times normal
* Alkaline phosphatase less than 2.5 times normal

Renal

* Creatinine less than 1.5 times upper limit of normal (ULN) OR
* BUN less than 1.5 times ULN

Cardiovascular

* No deep vein thrombosis within the past 3 weeks (must be clinically stable)

Pulmonary

* No pulmonary embolism within the past 3 weeks (must be clinically stable)

Other

* No peripheral neuropathy grade 2 or greater
* No active infection
* No other serious concurrent medical illness
* No concurrent illness that may obscure toxicity or dangerously alter drug metabolism
* No other malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* Must participate in the System for Thalidomide Education and Prescribing Safety program
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of effective contraception for 1 month before, during, and for 1 month after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior oral thalidomide or celecoxib for more than 2 months duration

Chemotherapy

* No prior oral etoposide or cyclophosphamide for more than 2 months duration
* Prior standard-dose IV etoposide and cyclophosphamide allowed

Endocrine therapy

* See Disease Characteristics
* Concurrent steroids allowed

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

Surgery

* See Disease Characteristics
* Prior surgery for relapsed or refractory disease allowed
* Recovered from prior surgery
* No concurrent surgery

Other

* No other concurrent investigational agents or treatment
* No other concurrent anticancer therapy
* Concurrent antiseizure medications allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-03 (Actual); Primary Completion 2005-08 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y. Wen, MD, Study Chair — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No